CLINICAL TRIAL: NCT01691937
Title: Continuous Right Thoracic Paravertebral Block on Postoperative Pain After Right Lobe Hepatectomy
Brief Title: Continuous Paravertebral Block on Postoperative Pain After Hepatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Principal Investigator, Wei Mei, Associate Prof., Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJMZK20120302
Record Dates: First submitted 2012-09-18; First posted 2012-09-25 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Right Lobe Hepatectomy
Keywords: Thoracic paravertebral block; Postoperative pain; Right lobe hepatectomy; Patient controlled analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Analgesia, Patient-Controlled; Sufentanil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PVB + PCA (Experimental): Continuous Paravertebral block with ropivacaine and Patient-controlled analgesia with sufentanil
  Interventions: Procedure: Continuous Paravertebral block with ropivacaine; Procedure: Patient-controlled analgesia with sufentanil
- Placebo PVB + PCA (Placebo Comparator): Continuous Paravertebral Block with Saline and Patient-controlled analgesia with sufentanil
  Interventions: Procedure: Patient-controlled analgesia with sufentanil; Procedure: Continuous Paravertebral Block with Saline

INTERVENTIONS:
Procedure: Continuous Paravertebral block with ropivacaine — Before anesthesia, continuous right thoracic paravertebral block of T7 is performed. After injection of 5 mL normal saline, a catheter (PAJUNK, Geisingen, Germany) is advanced medially the estimated distance to the paravertebral space. After injection of 1% lidocaine 15ml, the block level is tested by pinprick and recorded 15 minutes later. At the end of operation, syringe contained 0.2% ropivacaine is connected to paravertebral catheter, a 10ml bolus of 0.2% ropivacaine is injected via the paravertebral catheter, followed by an infusion of ropivacaine 0.2% at 6 ml/h for postoperative pain management.
  Arms: PVB + PCA
Procedure: Patient-controlled analgesia with sufentanil — Once arrival at the PACU, all patients were placed on a postoperative analgesic regimen that included patient-controlled analgesia with intravenous sufentanil (bolus 1μg, lockout time 10 min) and tramadol 100 mg IV for severe pain (NRS 6-10).
Procedure: Continuous Paravertebral Block with Saline — Before anesthesia, continuous right thoracic paravertebral block of T7 is performed. After injection of 5 mL normal saline, a catheter (PAJUNK, Geisingen, Germany) is advanced medially the estimated distance to the paravertebral space. After injection of 1% lidocaine 15ml, the block level is tested by pinprick and recorded 15 minutes later. At the end of operation, syringe contained 0.9% saline is connected to paravertebral catheter, a 10ml bolus of 0.9% saline is injected via the paravertebral catheter, followed by an infusion of 0.9% saline at 6 ml/h for postoperative pain management.
  Arms: Placebo PVB + PCA

SUMMARY:
Patients often experience moderate to severe postoperative pain, especially during the first hours after hepatectomy. Systemic opioids given with patient-controlled analgesia has be used after hepatectomy in many medical center(Aubrun, Monsel et al. 2001; Aubrun, Salvi et al. 2005), but the analgesic effect can be limited and undesirable side effects may occur.

A case report described that right thoracic paravertebral block reduced pain and analgesic requirements after right lobe hepatectomy(Ho, Karmakar et al. 2004). Compared with epidural analgesia, thoracic paravertebral block probably carries a much lower risk of spinal haematoma in the presence of moderate haemostatic deficiencies (Richardson and Lonnqvist 1998; Karmakar 2001).

We therefore designed a prospective, randomized, subject and assessor blinded, parallel-group, placebo controlled study to test the hypothesis that continuous right thoracic paravertebral analgesia decreases opioid consumption during the first 24 h after right lobe hepatectomy in patients receiving i.v. patient-controlled analgesia (PCA) with sufentanil.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 yrs
* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Undergo right lobe hepatectomy
* Informed consent

Exclusion Criteria:

* A known allergy to the drugs being used
* Coagulopathy, on anticoagulants
* Analgesics intake, history of substance abuse
* Participating in the investigation of another experimental agent
* Inability to properly describe postoperative pain to investigators (eg, language barrier, neuropsychiatric disorder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The cumulative opioid consumption | At 24 postoperative hours

SECONDARY OUTCOMES:
The pain scores determined by the numeric rating scale (NRS, 0-10) | At 1, 4, 8, 16, and 24 hrs after the surgery
Incidence of postoperative nausea and vomiting | Up to 24 postoperative hrs
Incidence of postoperative respiratory depression | Up to 24 postoperative hrs
Intraoperative bleeding | Up to 4 hours
Postoperative hospital length of stay | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, MD., Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Chen H, Liao Z, Fang Y, Niu B, Chen A, Cao F, Mei W, Tian Y. Continuous right thoracic paravertebral block following bolus initiation reduced postoperative pain after right-lobe hepatectomy: a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2014 Nov-Dec;39(6):506-12. doi: 10.1097/AAP.0000000000000167. PMID 25304475